CLINICAL TRIAL: NCT02075411
Title: A Randomized, Controlled Trial to Evaluate Opioid Usage Associated With Femoral Continuous Perineural Infusion and Femoral Single Shot Peripheral Nerve Block After a Hamstring Autograft Anterior Cruciate Ligament Repair.
Brief Title: Opioid Use in Single Shot Nerve Block vs Continuous Peripheral Nerve Infusion in Anterior Cruciate Ligament (ACL) Repair
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficult to enroll, parents/subjects prefer to choose type of anesthetic block.
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-009320
Record Dates: First submitted 2014-02-25; First posted 2014-03-03 (Estimated); Results first posted 2016-05-18 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-04

CONDITIONS: Injury of Anterior Cruciate Ligament
Keywords: anterior cruciate ligament reconstruction; transplantation allografts; adolescent; nerve block; pain
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Pain | interventions — Bupivacaine; Analgesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Males Single shot peripheral nerve block (Active Comparator): a single injection peripheral nerve block (FS/SS) of the femoral and sciatic nerves, Femoral Block - 0.25% bupivacaine (0.5 ml/kg, max 40 ml). The sciatic block will be performed using 0.125% bupivacaine (0.5 ml/kg, max 20 ml).
  Interventions: Drug: bupivacaine
- Females Single shot peripheral nerve block (Active Comparator): a single injection peripheral nerve block (FS/SS) of the femoral and sciatic nerves, Femoral Block - 0.25% bupivacaine (0.5 ml/kg, max 40 ml). The sciatic block will be performed using 0.125% bupivacaine (0.5 ml/kg, max 20 ml).
  Interventions: Drug: bupivacaine
- Males Continuous peripheral neural infusion (Active Comparator): The placement of a femoral continuous peripheral nerve infusion catheter (CPNI) and 0.25% bupivacaine (0.5 ml/kg, max 20 ml) will be injected under ultrasound guidance.
  Interventions: Device: continuous perineural infusion catheter
- Females Continuous peripheral neural infusion (Active Comparator): The placement of a femoral continuous peripheral nerve infusion catheter (CPNI) and 0.25% bupivacaine (0.5 ml/kg, max 20 ml) will be injected under ultrasound guidance.
  Interventions: Device: continuous perineural infusion catheter

INTERVENTIONS:
Drug: bupivacaine — Adolescent males receive the single shot femoral and sciatic nerve blocks prior to ACL repair.
  Males Single shot peripheral nerve block
  Other Names: sciatic nerve block; ACL repair
  Arms: Males Single shot peripheral nerve block
Drug: bupivacaine — Adolescent females receive the single shot femoral and sciatic nerve blocks prior to ACL repair.
  Females Single shot peripheral nerve block
  Other Names: sciatic nerve block; ACL repair
  Arms: Females Single shot peripheral nerve block
Device: continuous perineural infusion catheter — Adolescent males receive the continuous peripheral nerve block infusion catheter prior to ACL repair.
  Other Names: continuous peripheral nerve catheter infusion; pain control; ACL repair
  Arms: Males Continuous peripheral neural infusion
Device: continuous perineural infusion catheter — Adolescent females receive the continuous peripheral nerve block infusion catheter prior to ACL repair.
  Other Names: continuous peripheral nerve catheter infusion; pain control; ACL repair
  Arms: Females Continuous peripheral neural infusion

SUMMARY:
Anterior cruciate ligament repair using hamstring autograft in children is a painful orthopedic procedure. The current practice to provide analgesia for this procedure include femoral continuous perineural infusion and femoral single shot peripheral nerve block, along with perioperative opioids and NSAIDS both IV and orally. Since the use of opioids can be associated with adverse side effects, which include, but are not limited to nausea, vomiting, constipation, pruritus and respiratory depression, comparing the amount of opioid used with either analgesia delivery method is needed.

DETAILED DESCRIPTION:
The trial design is a prospective, randomized, open-label controlled, study. It is not possible to blind the treatment since a catheter must be left in place for the continuous infusion group.

Subjects will be randomized to either the femoral shot/continuous peripheral neural infusion FS-CPNI group or femoral shot/sciatic single shot FS-SS group. After induction of general anesthesia, subjects will receive either a single shot or continuous nerve block. The protocol will not dictate the conduct of the general anesthetic.

In the postoperative period, in addition to the standard monitoring in the recovery room, the numerical rating pain scale(NRS) scores of the patient will be recorded. The timing of the first rescue pain medication and total postoperative opioid and other analgesic medication administered during the hospital stay will be recorded. The patients will be followed in the hospital on the day of surgery (DOS) postoperatively until they are discharged home.

After discharge the patients will be contacted by phone and/or email postoperatively on a daily basis for 72 hours to collect information regarding their use of pain medications (timing and dose), quality of analgesia based on the NRS pain scale, and incidence of side effects. If patients need to be admitted to the hospital postoperatively, their opioid use, pain scores and complications will be recorded while in the hospital.

All the patients will be evaluated in the orthopedic clinic at two weeks, six weeks and six months to assess long term functional outcomes, pain scores and any signs of postoperative neurological deficits.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) physical status 1 or 2
* Male or female subjects ages 14 to 18 years old at time of procedure
* Patients who undergo an ACL repair using the hamstring autograft at The Children's Hospital of Philadelphia
* Parental/guardian permission (informed consent) and if appropriate, child assent

Exclusion Criteria:

* Parents/patients refusal to the placement of a femoral and/or sciatic nerve block
* Contraindications to femoral and/or sciatic nerve block:

  1. Infection
  2. Neurologic deficits, including motor and/or sensory deficit of the femoral and sciatic nerves.
* Patients' inability to participate in pain scoring because of developmental delay.
* Performance of an all-epiphyseal ACL repair.
* Allergy to any of the medications used in the study.
* Presence of a coagulopathy

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2014-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harshad Gurnaney, MBBS, MPH, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital Of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Beginning in June 2014, 49 potentially eligible patients were identified. Of these, 35 patients did not meet inclusion/exclusion criteria including, and 3 patients were unable to be contacted by phone pre-operatively. Of the remaining 11 potential patients, 10 declined study participation and only 1 signed consent to participate.
Pre-assignment Details: Only 1 subject signed consent to participate.
Groups:
- Males Single Shot Peripheral Nerve Block: a single injection peripheral nerve block (FS/SS) of the femoral and sciatic nerves, Femoral Block - 0.25% bupivacaine (0.5 ml/kg, max 40 ml). The sciatic block will be performed using 0.125% bupivacaine (0.5 ml/kg, max 20 ml).
  bupivacaine: Adolescent males receive the single shot femoral and sciatic nerve blocks prior to ACL repair.
  Males Single shot peripheral nerve block
- Females Single Shot Peripheral Nerve Block: a single injection peripheral nerve block (FS/SS) of the femoral and sciatic nerves, Femoral Block - 0.25% bupivacaine (0.5 ml/kg, max 40 ml). The sciatic block will be performed using 0.125% bupivacaine (0.5 ml/kg, max 20 ml).
  bupivacaine: Adolescent females receive the single shot femoral and sciatic nerve blocks prior to ACL repair.
  Females Single shot peripheral nerve block
Period: Overall Study
Arm/Group | Males Single Shot Peripheral Nerve Block | Females Single Shot Peripheral Nerve Block | Males Continuous Peripheral Neural Infusion | Females Continuous Peripheral Neural Infusion
Started | 0 | 0 | 0 | 1
Completed | 0 | 0 | 0 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Males Single Shot Peripheral Nerve Block | Females Single Shot Peripheral Nerve Block | Males Continuous Peripheral Neural Infusion | Females Continuous Peripheral Neural Infusion | Total
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 1
Age, Categorical [Number; unit: participants]
  <=18 years |  |  |  | 1 | 1
  Between 18 and 65 years |  |  |  | 0 | 0
  >=65 years |  |  |  | 0 | 0
Gender [Number; unit: participants]
  Female |  |  |  | 1 | 1
  Male |  |  |  | 0 | 0
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native |  |  |  | 0 | 0
  Asian |  |  |  | 0 | 0
  Native Hawaiian or Other Pacific Islander |  |  |  | 0 | 0
  Black or African American |  |  |  | 0 | 0
  White |  |  |  | 1 | 1
  More than one race |  |  |  | 0 | 0
  Unknown or Not Reported |  |  |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  |  |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Opioid Pain Medication
Description: total postoperative opioid pain medication used during the first 72 hours after the procedure
Time Frame: 72 hours post-operatively
Population: Sample size was too small to conduct outcome analysis
Arm/Group | Males Single Shot Peripheral Nerve Block | Females Single Shot Peripheral Nerve Block | Males Continuous Peripheral Neural Infusion | Females Continuous Peripheral Neural Infusion
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Duration of Analgesia in the Single Injection Nerve Block and the Continuous Peripheral Neural Infusion Group
Description: Determine the duration of analgesia in the 2 groups. Analgesic duration will be the time interval between the end of the operation and the time of first administration of opioid for pain relief
Time Frame: 72 hours post-operatively
Population: Sample size was too small to conduct outcome analysis
Arm/Group | Males Single Shot Peripheral Nerve Block | Females Single Shot Peripheral Nerve Block | Males Continuous Peripheral Neural Infusion | Females Continuous Peripheral Neural Infusion
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Other Pre Specified Outcome: Failure of Nerve Block Procedures
Description: We will determine the proportion of failure of the nerve block procedures as assessed by absence of a sensory block in the distribution of the femoral or sciatic nerves. The analysis will be of the numerical rating scale (NRS) scores immediately on arrival (baseline) in the recovery room and then every 6 hours over the first 72 hours post-op in the 2 groups.
Time Frame: 72 hours post-operatively
Population: Sample size was too small to conduct outcome analysis
Arm/Group | Males Single Shot Peripheral Nerve Block | Females Single Shot Peripheral Nerve Block | Males Continuous Peripheral Neural Infusion | Females Continuous Peripheral Neural Infusion
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 72 hours post-operatively
Arm/Group | Males Single Shot Peripheral Nerve Block | Females Single Shot Peripheral Nerve Block | Males Continuous Peripheral Neural Infusion | Females Continuous Peripheral Neural Infusion
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
Due limited enrollment and early termination of this study, analysis of outcome data was not possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes